CLINICAL TRIAL: NCT04524403
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Miricorilant in Obese Adult Patients With Schizophrenia Taking Antipsychotic Medications (GRATITUDE II)
Brief Title: A Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Miricorilant in Obese Adult Patients With Schizophrenia While Taking Antipsychotic Medications (GRATITUDE II)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CORT118335-877
Record Dates: First submitted 2020-08-06; First posted 2020-08-24 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Antipsychotic-induced Weight Gain (AIWG)
Keywords: Antipsychotic-induced weight gain (AIWG); Obesity; Weight Gain; Mental disorders; Schizophrenia; Risperidone; Paliperidone; Quetiapine; Olanzapine
MeSH Terms: conditions — Obesity; Weight Gain; Mental Disorders; Schizophrenia | interventions — CORT118335

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Miricorlilant 600 mg (Experimental): Patients who meet the entry criteria will be randomized to receive 600 mg miricorilant for 26 weeks.
  Interventions: Drug: Miricorlilant
- Miricorlilant 900 mg (Experimental): Patients who meet the entry criteria will be randomized to receive 900 mg miricorilant for 26 weeks.
  Interventions: Drug: Miricorlilant
- Placebo (Placebo Comparator): Patients who meet the entry criteria will be randomized to receive placebo for 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Miricorlilant — Miricorilant 600 mg (4 X 150 mg) for once-daily for oral dosing
  Other Names: CORT118335
  Arms: Miricorlilant 600 mg
Drug: Miricorlilant — Miricorilant 900 mg (6 X 150 mg) for once-daily for oral dosing
  Other Names: CORT118335
  Arms: Miricorlilant 900 mg
Drug: Placebo — Placebo for once-daily oral dosing
  Arms: Placebo

SUMMARY:
This Phase 2, double-blind, placebo-controlled, randomized study is to assess the safety, efficacy, and pharmacokinetics (PK) of miricorilant (CORT118335) in obese patients with schizophrenia treated with antipsychotic medications.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study that will assess the safety, efficacy, and PK of miricorilant in obese patients with schizophrenia who are currently taking olanzapine, risperidone, paliperidone, or quetiapine.

Patients who meet the criteria for the Study CORT118335-877 will be randomized on Day 1 to receive 600 mg miricorilant, 900 mg miricorilant, or placebo for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of schizophrenia
* Are currently taking olanzapine, risperidone, paliperidone, or quetiapine and have gained weight from treatment while on these medications
* Must be on a stable dose of medication for 1 month prior to Screening
* Have a BMI ≥30 kg/m^2.

Exclusion Criteria:

* Have a history of a medical condition affecting body weight (eg, poorly controlled hyper- or hypothyroidism; eating disorder such as anorexia, bulimia, or binge eating; or polycystic ovary syndrome)
* Have poorly controlled diabetes mellitus
* Have poorly controlled hypertension
* Have a history of symptomatic hypotension
* Have a history of orthostatic hypotension
* Have a history of a seizure disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Juneja, MD, Study Director — Corcept Therapeutics
Locations (39):
- United States (39):
  - Site #143, Bentonville, Arkansas
  - Site # 249, Little Rock, Arkansas
  - Site #153, Culver City, California
  - Site #239, Garden Grove, California
  - Site # 243, Glendale, California
  - Site #134, Lemon Grove, California
  - Site #163, Oceanside, California
  - Site # 247, Pico Rivera, California
  - Site # 229, Rancho Cucamonga, California
  - Site # 237, San Diego, California
  - Site # 150, Stanford, California
  - Site #202, Miami, Florida
  - Site #144, Miami Lakes, Florida
  - Site #144, North Miami, Florida
  - Site #241, Okeechobee, Florida
  - Site # 240, Chicago, Illinois
  - Site #140, Chicago, Illinois
  - Site #140, Lincolnwood, Illinois
  - Site #225, Flowood, Mississippi
  - Site #224, St Louis, Missouri
  - Site #217, Lincoln, Nebraska
  - Site #151, Las Vegas, Nevada
  - Site # 244, Cedarhurst, New York
  - Site #216, New York, New York
  - Site # 245, New York, New York
  - Site #231, Staten Island, New York
  - Site # 248, Charlotte, North Carolina
  - Site #181, Raleigh, North Carolina
  - Site # 181, Raleigh, North Carolina
  - Site #107, Dayton, Ohio
  - Site # 230, North Canton, Ohio
  - Site #166, Philadelphia, Pennsylvania
  - Site #235, Thorndale, Pennsylvania
  - Site #235, West Chester, Pennsylvania
  - Site #223, Austin, Texas
  - Site #206, DeSoto, Texas
  - Site #066, Houston, Texas
  - Site #165, Richardson, Texas
  - Site #137, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Miricorlilant 600 mg: Patients who meet the entry criteria will be randomized to receive 600 mg miricorilant for 26 weeks.
  Miricorlilant: Miricorilant 600 mg (4 X 150 mg) tablets for once-daily oral dosing
- Miricorlilant 900 mg: Patients who meet the entry criteria will be randomized to receive 900 mg miricorilant for 26 weeks.
  Miricorlilant: Miricorilant 900 mg (6 X 150 mg) tablets for once-daily oral dosing
Period: Overall Study
Arm/Group | Miricorlilant 600 mg | Miricorlilant 900 mg | Placebo
Started | 50 | 48 | 52
Completed | 33 | 37 | 34
Not Completed | 17 | 11 | 18
Not completed — Withdrawal by Subject | 10 | 3 | 8
Not completed — Lost to Follow-up | 3 | 4 | 3
Not completed — Adverse Event | 3 | 1 | 4
Not completed — Non-compliant with study drug | 1 | 2 | 3
Not completed — Moved | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Miricorlilant 600 mg | Miricorlilant 900 mg | Placebo | Total
Number analyzed (Participants) | 50 | 48 | 52 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (10.80) | 46.4 (10.88) | 47.5 (10.27) | 46.5 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 18 | 54
  Male | 33 | 29 | 34 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 4 | 21
  Not Hispanic or Latino | 40 | 40 | 48 | 128
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 28 | 29 | 28 | 85
  White | 19 | 17 | 21 | 57
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 50 | 48 | 52 | 150
Body weight [Mean (Standard Deviation); unit: kg] | 115.41 (24.24) | 108.02 (19.78) | 118.11 (25.71) | 113.98 (23.69)
Waist-to-hip ratio [Mean (Standard Deviation); unit: Ratio] | 0.991 (0.07) | 0.999 (0.06) | 0.992 (0.08) | 0.994 (0.07)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body Weight
Time Frame: Baseline Day 1 and Week 26
Population: The Efficacy Evaluable Population was patients who received ≥4 weeks of study drug and had body weight measurements at Baseline and on Week 26.
Measure: Least Squares Mean (Standard Error); unit: kg
Groups:
- Placebo: Patients who meet the entry criteria will be randomized to receive placebo once daily for 26 weeks.
  Placebo: Placebo for oral dosing
Arm/Group | Miricorlilant 600 mg | Miricorlilant 900 mg | Placebo
Number analyzed (Participants) | 37 | 39 | 35
kg | -1.41 (0.644) | -0.91 (0.631) | -1.66 (0.644)
Statistical Analysis 1: Comparison: Miricorlilant 600 mg vs Placebo; Test type: Superiority; p = 0.7870, Mixed Models Analysis; Least Squares Mean Difference = 0.24, 95% CI 2-sided [-1.52 to 2.01]
Statistical Analysis 2: Comparison: Miricorlilant 900 mg vs Placebo; Test type: Superiority; p = 0.4018, Mixed Models Analysis; Least Squares Mean Difference = 0.75, 95% CI 2-sided [-1.01 to 2.51]

2. Secondary Outcome: Change From Baseline in Body Weight for Both Dose Levels of Miricorilant Combined Versus Placebo
Time Frame: Baseline Day 1 and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Groups:
- Miricorilant 600 mg or 900 mg: Patients who meet the entry criteria will be randomized to receive miricorilant 600 mg (4 X 150 mg) tablets or 900 mg (6 X 150 mg) tablets orally once-daily for 26 weeks.
- Placebo: Patients who meet the entry criteria will be randomized to receive placebo once daily for 26 weeks.
Arm/Group | Miricorilant 600 mg or 900 mg | Placebo
Number analyzed (Participants) | 76 | 35
kg | -1.16 (0.454) | -1.65 (0.642)
Statistical Analysis 1: Comparison: Miricorilant 600 mg or 900 mg vs Placebo; Test type: Superiority; p = 0.5228, Mixed Models Analysis; Least Squares Mean Difference = 0.50, 95% CI 2-sided [-1.03 to 2.02]

3. Secondary Outcome: Percentage of Patients Achieving a ≥5% Weight Loss for Miricorilant Versus Placebo
Description: Percentage of patients achieving a ≥5% weight loss for 600 mg miricorilant versus placebo and 900 mg miricorilant versus placebo
Time Frame: Baseline Day 1 to Week 26
Population: The Efficacy Evaluable Population was patients who received ≥4 weeks of study drug and had Baseline and ≥1 body weight measurement on or after Week 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Miricorlilant 600 mg | Miricorlilant 900 mg | Placebo
Number analyzed (Participants) | 45 | 46 | 48
Participants | 12 | 7 | 8
Statistical Analysis 1: Comparison: Miricorlilant 600 mg vs Placebo; Test type: Superiority; p = 0.2537, Regression, Logistic; Odds Ratio (OR) = 1.781, 95% CI 2-sided [0.661 to 4.802]
Statistical Analysis 2: Comparison: Miricorlilant 900 mg vs Placebo; Test type: Superiority; p = 0.8740, Regression, Logistic; Odds Ratio (OR) = 0.916, 95% CI 2-sided [0.308 to 2.722]

4. Secondary Outcome: Change From Baseline in Waist-to-hip Ratio for Miricorilant Versus Placebo
Time Frame: Baseline Day 1 and Week 26
Population: The Efficacy Evaluable Population was patients who received ≥4 weeks of study drug and had weight and hip measurements at Baseline and on Week 26.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Miricorlilant 600 mg | Miricorlilant 900 mg | Placebo
Number analyzed (Participants) | 37 | 39 | 35
Ratio | 0.002 (0.0077) | 0.009 (0.0075) | 0.002 (0.0077)
Statistical Analysis 1: Comparison: Miricorlilant 600 mg vs Placebo; Test type: Superiority; p = 0.9870, Mixed Models Analysis; Least Squares Mean Difference = 0.000, 95% CI 2-sided [-0.021 to 0.021]
Statistical Analysis 2: Comparison: Miricorlilant 900 mg vs Placebo; Test type: Superiority; p = 0.4624, Mixed Models Analysis; Least Squares Mean Difference = 0.008, 95% CI 2-sided [-0.013 to 0.029]

5. Other Pre Specified Outcome: Number of Patients With One or More Treatment-emergent Adverse Events
Time Frame: Baseline Day 1 to Week 30
Population: The Safety Population was patients who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Miricorlilant 600 mg | Miricorlilant 900 mg | Placebo
Number analyzed (Participants) | 50 | 48 | 52
Participants | 26 | 21 | 21

6. Other Pre Specified Outcome: Number of Patients With One or More Treatment-emergent Serious Adverse Events
Time Frame: Baseline Day 1 to Week 30
Population: The Safety Population was patients who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Miricorlilant 600 mg | Miricorlilant 900 mg | Placebo
Number analyzed (Participants) | 50 | 48 | 52
Participants | 1 | 2 | 2

7. Other Pre Specified Outcome: Number of Patients With One or More Treatment-emergent Adverse Events Leading to Study Drug Discontinuation
Time Frame: Baseline Day 1 to Week 30
Population: The Safety Population was patients who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Miricorlilant 600 mg | Miricorlilant 900 mg | Placebo
Number analyzed (Participants) | 50 | 48 | 52
Participants | 7 | 5 | 4

ADVERSE EVENTS:
Time Frame: Baseline Day 1 to Week 30
Description: The Safety Population was patients who received ≥1 dose of study drug.
Arm/Group | Miricorlilant 600 mg | Miricorlilant 900 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/48 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/50 | 2/48 | 2/52
Other Adverse Events (participants affected / at risk) | 8/50 | 3/48 | 4/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Miricorlilant 600 mg (N=50) | Miricorlilant 900 mg (N=48) | Placebo (N=52)
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Regressive behavior (Psychiatric disorders) | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Miricorlilant 600 mg (N=50) | Miricorlilant 900 mg (N=48) | Placebo (N=52)
Alanine aminotransferase increased (Investigations) | 4 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 0
Headache (Nervous system disorders) | 4 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual publications will be allowed before publication of the multicenter results, except as agreed with the Sponsor. The Investigator agrees to submit all manuscripts or abstracts to the Sponsor for review before submission to the publisher.

DOCUMENTS (2):
  • Study Protocol (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT04524403/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT04524403/SAP_001.pdf